CLINICAL TRIAL: NCT04299698
Title: Interaction of Genetic and Environmental Factors for Body Fat Mass Control: Observational Study for Lifestyle Modification and Genotyping
Brief Title: Interaction of Genetic and Environmental Factors for Body Fat Mass Control
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Semiconductor R&D center (Unknown)
Responsible Party: Principal Investigator, Woong-Yang Park, Head of Samsung Genomic institute, Samsung Medical Center
Other Study IDs: 2017-03-064
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Unrecognized Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Carbohydrate reduction group: Participants chose to control their body fat mass by reducing their carbohydrate intake through observation study periods.
  Interventions: Behavioral: lifestyle
- Fat reduction group: Participants chose to control their body fat mass by reducing their fat intake through observation study periods.
  Interventions: Behavioral: lifestyle
- Intense exercise group: Participants chose to control their body fat mass by vigorously increasing the time and intensity of exercise through observation study periods.
  Interventions: Behavioral: lifestyle
- Moderate exercise group: Participants chose to control their body fat mass by moderately increasing the time and intensity of exercise through observation study periods.
  Interventions: Behavioral: lifestyle

INTERVENTIONS:
Behavioral: lifestyle — Participants who desire to control body fat mass chose the one of lifestyle modification on their diet or exercise.

SUMMARY:
Although the effect of interaction between genetic and environmental factors on body fat mass (BFM) has been proposed, how lifestyle changes affect body weight with regard to the genetic composition needs to be verified. The investigators designed an observational study, consisting of healthy adults with single nucleotide polymorphism (SNP) genotyping and longitudinal monitoring of lifestyle including food consumption and physical activities. The investigators recruited the participants who desired to control their body fat mass. Participants freely choose one of the options among carbohydrate intake reduction, fat intake reduction or exercise amount increment to control their body fat mass. Their lifelog on exercise and diet were collected, using a wearable device, for three months. Further, the investigators assessed anthropometric and serologic markers to measure the effect of participant's lifestyle modification. The investigators evaluate the influence of genetic compositions on body fat reduction induced by lifestyle change. Four different genome-wide polygenic scores (GPS) of volunteers are calculated to test the genetic effects of each modification. In this lifestyle observational study, the investigators expect to validate the interaction of genetic and environmental factors in determining BFM, and implicate the healthcare utility of lifestyle modifications using personalized and genomic perspective.

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 65

Exclusion Criteria:

* Among those reveal to participate one who is under diabetes condition were excluded on the study.
* Pregnant women
* Participants taking weight control pills

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are all lived in South Korea in Seoul and Kyeonggi-do.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Change of body fat mass | baseline and 14 weeks
  Anthropometric data including body fat mass were measured by InBody720 --assessing whole and segmental body composition.

CONTACTS AND LOCATIONS:
Overall Officials: Woong-Yang Park, MD, Study Chair — Samsung Genomic Institute
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
A plan is undecided yet.